CLINICAL TRIAL: NCT00772057
Title: Early Primary Prophylaxis With Beta-Blockers In Prevention Of Growth Of Small Esophageal Varices In Cirrhosis: A Randomized Controlled Trial
Brief Title: Beta-blockers for Prevention Of Growth Of Small Esophageal Varices In Cirrhosis: An Randomized Controlled Trial (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr S K Sarin, Department of Gastroenterology, G B Pant Hospital, New Delhi, India
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2008-PHT-02
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2008-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol group (Active Comparator)
  Interventions: Drug: Propranolol
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Beta-blocker (propranolol) was started at a dose of 20 mg twice daily. The principle of incremental dosing was used to achieve the target heart rate for propranolol. The dose was increased every alternate day to achieve a target heart rate of 55/min or to the maximal dose to 360 mg/day if the medication was well tolerated and the systolic blood pressure was >90 mm Hg. On the occurrence of intolerable adverse effects, systolic blood pressure <90 mm Hg or pulse rate <55/min, the dose of the medication was decreased step-wise, and eventually stopped if these adverse events persisted. Reintroduction of the medication was attempted if cessation of the medication did not result in improvement of the reported side-effect.
  Arms: Propranolol group
Drug: Placebo — Placebo tablets given two times daily.
  Arms: Placebo group

SUMMARY:
Background and Aims: The efficacy of portal pressure reduction by beta blockers for the management of small (≤5 mm) esophageal varices in patients of cirrhosis is not clear. The present randomized controlled trial aims to address these issues. The investigators also assessed the utility of serial HVPG measurements in these patients.

Patients and Methods: Consecutive patients with cirrhosis with small varices, with no history of variceal bleed, were randomized to receive propranolol or placebo. These patients were further randomized to undergo no HVPG, only baseline HVPG, or serial HVPG measurement. Propranolol was titrated to reduce heart-rate to 55/min.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis was made
* Age was between 18 and 70 years
* Esophageal varices were small (i.e. ≤5 mm or of grade 1 or 2 according to Conn et al).

Exclusion Criteria:

* Presence of previous variceal bleeding
* Previous medical, surgical or endoscopic treatment for portal hypertension
* Child-Pugh score >13
* Neoplastic disease of any site
* Splenic or portal vein thrombosis
* Concurrent illnesses expected to decrease life expectancy to less than one year
* Pregnancy
* Contraindication to beta-blockers (atrioventricular block, sinus bradycardia with heart rate <50 beats per minute, arterial hypotension with systolic blood pressure <90 mm Hg, heart failure, asthma, peripheral arterial disease, or diabetes needing insulin treatment)
* Concurrent anti-viral treatment during the study period
* Inability to perform follow-up
* Failure to give consent to participate in the study.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study was the development of large (>5 mm) esophageal varices (grade 3 or 4 by Conn's classification) | 24 months

SECONDARY OUTCOMES:
Secondary endpoints were variceal bleeding, death, adverse effects of beta blockers, and hemodynamic response to beta-blocker in patients who underwent serial HVPG | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — G B Pant Hospital
Locations (1):
- Department of Gastroenterology, G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India